CLINICAL TRIAL: NCT05266963
Title: Pancreatic Enzyme Replacement and Glucose Regulation in Type 1 Diabetes
Acronym: CREON
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Moore, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210734
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancrelipase

STUDY DESIGN:
Intervention Model Description: Participants will receive CREON and placebo in a random, blinded order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CREON (Active Comparator): CREON is a pancreatic enzyme replacement
  Interventions: Drug: CREON
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CREON — The study will enroll 6-10 adult subjects with T1D who will receive both pancreatic enzyme replacement (CREON) or placebo each for 7 days in a random order. The effect of the intervention will be monitored by continuous glucose monitoring, diet recording, capsule counts, a mixed-meal tolerance test, and a survey to assess symptoms of PEI. This study design will allow for estimation of the effect of pancreatic enzyme replacement on the measured parameters.
  Arms: CREON
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Recent studies have demonstrated reduced pancreatic volume is present within months of T1D diagnosis in children, adolescents, and adults. As the pancreatic beta cells constitute only 1-2% of the pancreas, the degree of reduction in pancreas volume at disease onset suggests exocrine involvement, challenging the established paradigm of T1D being solely a disease of the endocrine pancreas.

To date there has not been an investigation of the potential for pancreatic enzyme replacement therapy in the management of T1D. In individuals with cystic fibrosis-related diabetes, enzyme replacement has been shown to reduce post-prandial glycemia excursions, which are reflected in improved GLP-1 responses to mixed meal tolerance testing. As post-prandial excursions and glucose variability are a significant challenge in T1D, how enzyme replacement may impact these parameters is an important question.

The investigators hypothesize that patients with T1DM who have reduced pancreatic volume will have improved glycemic responsiveness, reduced hypoglycemia, and improved symptoms of pancreatic exocrine insufficiency when treated with pancreatic enzyme replacement (CREON).

ELIGIBILITY:
Inclusion Criteria:

* Currently receive care at the Eskind Diabetes Clinic at Vanderbilt University Medical Center
* Diagnosed with T1DM for at least 12 months
* Age over 18
* Total daily dose of insulin greater than 0.7u/kg/day
* Current use of a continuous glucose monitor
* Current use of smart phone
* Able to read and speak English
* Willingness and ability to download and provide CGM and pump (if applicable) data
* Reduction of pancreas volume (<0.6mL/kg body weight)

Exclusion Criteria:

* History of celiac disease or inflammatory bowel disease
* Use of medication or supplements other than insulin to control blood glucose
* Pregnancy or breast feeding
* Following a restrictive diet (such as very low carb diet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share PHI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Vanderbilt University Medical Center from September 2022 through March 2024. Subjects were eligible based on reduced pancreas volume as determined through their prior participation in MAP-T1D (IRB 130833).
Pre-assignment Details: Eleven (11) participants were enrolled to achieve completion goal of ten (10). One subject withdrew at end of drug period A due to failed OGTT and unwillingness to continue.
Groups:
- CREON, Then Placebo; Placebo, Then CREON: CREON is a pancreatic enzyme replacement
  CREON: The study will enroll 6-10 adult subjects with T1D who will receive both pancreatic enzyme replacement (CREON) or placebo each for 7 days in a random order. The effect of the intervention will be monitored by continuous glucose monitoring, diet recording, capsule counts, a mixed-meal tolerance test, and a survey to assess symptoms of PEI. This study design will allow for estimation of the effect of pancreatic enzyme replacement on the measured parameters.
Period: Drug Period A
Arm/Group | CREON, Then Placebo | Placebo, Then CREON
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout
Arm/Group | CREON, Then Placebo | Placebo, Then CREON
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Drug Period B (Crossover)
Arm/Group | CREON, Then Placebo | Placebo, Then CREON
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Although 11 participants were enrolled, only 10 completed both treatment periods, so those 10 are the only ones included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | CREON, Then Placebo | Placebo, Then CREON | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 44.2 [22.7 to 72.2] | 22.3 [18.1 to 32.3] | 33.3 [18.1 to 72.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Weight [Mean (Full Range); unit: kg] | 69.7 [61.2 to 75.7] | 84.8 [68.3 to 118.7] | 77.3 [61.2 to 118.7]
Pancreatic exocrine insufficiency score [Mean (Full Range); unit: units on a scale] — We will use the pancreatic exocrine insufficiency questionnaire (PEI-Q) to quantitate symptoms of PEI and their relative change from baseline to after treatment with placebo and Creon in a random order. Minimum score is 0, and maximum score is 4. Higher scores correlate to worse outcome, i.e., increased abdominal symptoms and bowel movement symptoms.
  units on a scale | 0.44 [0.143 to 0.821] | 0.312 [0 to 0.833] | 0.376 [0 to 0.833]
C-peptide AUC [Mean (Full Range); unit: ng*hr/mL] | 44.4 [19.7 to 128.8] | 24.9 [17.1 to 39.4] | 34.4 [17.1 to 128.8]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Glucose Regulation
Description: Mixed meal tolerance testing (MMTT) will be used to assess glucose regulation via c-peptide AUC at baseline, and after treatment with placebo and CREON in a random order.
Time Frame: through study completion (4-5 weeks)
Population: This analysis population is the 10 participants who completed both drug periods of the study. Five received CREON, then placebo, and the other five received placebo, then CREON.
Measure: Mean (Full Range); unit: ng*hr/mL
Groups:
- Placebo: CREON is a pancreatic enzyme replacement
  CREON: The study will enroll 6-10 adult subjects with T1D who will receive both pancreatic enzyme replacement (CREON) or placebo each for 7 days in a random order. The effect of the intervention will be monitored by continuous glucose monitoring, diet recording, capsule counts, a mixed-meal tolerance test, and a survey to assess symptoms of PEI. This study design will allow for estimation of the effect of pancreatic enzyme replacement on the measured parameters.
Arm/Group | CREON | Placebo
Number analyzed (Participants) | 10 | 10
ng*hr/mL
  Baseline | 34.42 [17.1 to 128.8] | 34.42 [17.1 to 128.8]
  End of Drug Period | 35.44 [19.14 to 125.7] | 39.03 [15.95 to 160.48]
Statistical Analysis 1: Comparison: CREON vs Placebo; Test type: Superiority — Statistical analysis will be performed using a paired samples Wilcoxon test to compare differences between the two groups; p = 0.43, Wilcoxon (Mann-Whitney); Wilcoxon matched-pairs

2. Primary Outcome: Patient-reported Change in Pancreatic Exocrine Insufficiency (PEI) Symptoms
Description: We will use the pancreatic exocrine insufficiency questionnaire (PEI-Q) to quantitate symptoms of PEI and their relative change from baseline to after treatment with placebo and Creon in a random order. Minimum score is 0, and maximum score is 4. Higher scores correlate to worse outcome, i.e., increased abdominal symptoms and bowel movement symptoms.
Time Frame: through study completion (4-5 weeks)
Population: This analysis population is the 10 participants who completed both drug periods of the study. Five participants received CREON, then placebo, and the other five received placebo, then CREON.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CREON | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 0.376 [0 to 0.833] | 0.376 [0 to 0.833]
  End of Drug Period | 0.382 [0 to 0.893] | 0.346 [0 to 0.81]
Statistical Analysis 1: Comparison: CREON vs Placebo; Test type: Superiority — Statistical analysis will be performed using a standard two-tailed t test to compare differences between the two groups; p = 0.52, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 1 month per participant.
Groups:
- Placebo: Placebo
  Placebo: The study will enroll 6-10 adult subjects with T1D who will receive both pancreatic enzyme replacement (CREON) or placebo each for 7 days in a random order.
Arm/Group | CREON | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The intervention was given for a relatively short time, most patients had significantly reduced pancreas volume, and most had long histories of T1D. The baseline C-peptide levels in the subjects were very low. Assessment in individuals with new onset T1D, in younger subjects, or in individuals with greater residual beta cell function could produce different results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05266963/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05266963/SAP_001.pdf
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT05266963/ICF_002.pdf